CLINICAL TRIAL: NCT03385655
Title: Prostate Cancer Biomarker Enrichment and Treatment Selection (PC-BETS) Study
Brief Title: Prostate Cancer Biomarker Enrichment and Treatment Selection
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Canadian Cancer Clinical Trials Network (Unknown); BC Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I234
Record Dates: First submitted 2017-12-12; First posted 2017-12-28 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — adavosertib; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine; darolutamide; 2-(3-(4-((2,6-dimethylmorpholino)methyl)styryl)-1H-indazol-6-yl)-5'-methoxyspiro(cyclopropane-1,3'-indolin)-2'-one; ipatasertib; durvalumab; tremelimumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- WEE-1 inhibitor - ARM CLOSED (Experimental)
  Interventions: Drug: Adavosertib
- cMET inhibitor (Experimental)
  Interventions: Drug: Savolitinib
- novel non-steroidal androgen receptor (AR) antagonist (Experimental)
  Interventions: Drug: Darolutamide
- CFI400945 PLK4 inhibitor - ARM CLOSED (Experimental)
  Interventions: Drug: CFI-400945
- Ipatasertib AKT inhibitor (Experimental)
  Interventions: Drug: Ipatasertib
- Durvalumab and Tremelimumab immunotherapy (Experimental)
  Interventions: Drug: Durvalumab and Tremelimumab
- Carboplatin platinum based chemotherapy (Experimental)
  Interventions: Drug: Carboplatin

INTERVENTIONS:
Drug: Adavosertib — 250mg, may dose escalate to 300mg if no drug-related GI tox in cycle 1
  Arms: WEE-1 inhibitor - ARM CLOSED
Drug: Savolitinib — 600mg once daily, orally.
  Arms: cMET inhibitor
Drug: Darolutamide — 600mg twice daily, orally.
  Arms: novel non-steroidal androgen receptor (AR) antagonist
Drug: CFI-400945 — Dose level assigned at enrollment, starting at 32mg/day on Days 1-7 and 15-21 or 15-28 depending on toxicity experienced.
  Arms: CFI400945 PLK4 inhibitor - ARM CLOSED
Drug: Ipatasertib — 400mg daily 3 weeks on, 1 week off
  Arms: Ipatasertib AKT inhibitor
Drug: Durvalumab and Tremelimumab — Durvalumab 1500mg day 1 every 4 weeks; Tremelimumab 225mg day 1 cycle 1
  Arms: Durvalumab and Tremelimumab immunotherapy
Drug: Carboplatin — AUC 5 IV 60min Day 1 q 21 days
  Arms: Carboplatin platinum based chemotherapy

SUMMARY:
The purpose of the pre-study screening is to test for DNA abnormalities or biomarkers.

DETAILED DESCRIPTION:
This testing will be done on a samples of blood to see whether or not patients are eligible to take part in one of the sub-studies. Each study will be looking at what effects a new drug or drugs has on prostate cancer and will also be looking at the side effects of treatment. The purpose of the main studies is to see if the biomarkers that were identified screening samples can help predict which patients are most likely to be helped by that drug or drugs and to see how the cancer cells respond to treatment.

ELIGIBILITY:
Inclusion Criteria:

The following will be required prior to REGISTRATION:

* Patients must have histologically confirmed adenocarcinoma of the prostate without pathologic or clinical evidence (e.g. PSA < 2.0 μg/L with liver metastases) of small cell neuroendocrine differentiation.
* Patients must consent prior to blood collection for screening correlative testing by a central reference laboratory. The screening blood sample cannot be sent for analysis prior to screening registration.
* All patients must have consented to the release of a tumour block from their primary or metastatic tumour. The centre/pathologist must have agreed to the submission of the specimen(s). Contact CCTG if no archival tissue is available.
* Patients must have evidence of castrate resistance with either biochemical or radiological disease progression in the setting of surgical or medical castration:

PSA Progression:

* Minimum of two rising PSA values from a baseline measurement with an interval of ≥ 1 week between each measurement
* PSA must be ≥ 2.0 µg/L (ng/mL)

Objective progression:

* RECIST 1.1, or
* PCWG3 Criteria for bone progression

Surgical/Medical Castration:

* Prior bilateral orchiectomy, or
* LHRH agonist/antagonist and testosterone < 50 ng/dL or < 1.7 nmol/L. LHRH agonist/antagonist therapy must be maintained for the duration of study therapy and if previously discontinued, must be restarted and castrate level of testosterone present.
* Patients must be ≥18 years of age.
* ECOG performance status 0 or 1 (Appendix I) and have a life expectancy of ≥ 6 months.
* Patients must have radiologically documented disease (measurable or non-measurable as defined by RECIST 1.1. Patients with elevated PSA only are not eligible.
* Neutrophils ≥ 1.5 x 10^9/L
* Platelets ≥ 100 x 10^9/L
* Hemoglobin ≥ 90 g/L; contact CCTG if hemoglobin is between 80-89 g/L, patient is not decompensated, is asymptomatic and transfusion is not indicated.
* Serum potassium within normal limits
* Bilirubin ≤ 1.5 ULN; if confirmed Gilbert's then bilirubin ≤ 3.0 x ULN
* ALT ≤ 2.5 x ULN; if patient has liver metastases ≤ 5.0 x ULN
* Serum creatinine ≤ 1.5 x ULN or Creatinine clearance ≥ 45 mL/min; measured directly by 24-hour urine sampling OR as calculated by Cockcroft and Gault equation: Males: GFR = 1.23 x (140-age) x weight in kg/serum creatinine in μmol/L
* Patient consent for screening and subsequent enrollment (as applicable) must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to screening and subsequent enrollment (as applicable) in the trial to document their willingness to participate.

Additional Criteria to be met prior to SUB-STUDY ENROLLMENT:

* Patients must have recovered from any treatment-related toxicities prior to enrollment (unless ≤ grade 1, irreversible, or considered by investigator as not clinically significant).
* Prior major surgery is permitted provided that a minimum of 14 days have elapsed between any major surgery and enrollment (7 days for minor surgery e.g. port insertion), and that wound healing has occurred.
* Prior external beam radiation or radium-223 is permitted provided a minimum of 28 days (4 weeks) have elapsed between the last dose and enrollment. Consult CCTG if patients have received other therapeutic radioisotopes. Exceptions may be made for low-dose non-myelosuppressive radiotherapy after consultation with CCTG. Concurrent radiation is not permitted. If radiation is required for example for pain control, it must be completed prior to enrollment. Prior strontium-89 at any time is not permitted.
* Previous Hormone Therapy: Patients must have received prior hormonal treatment with at least one of: abiraterone acetate, enzalutamide, apalutamide (ARN-509), darolutamide (ODM-201), TAK-700 and TOK-001 or other next-generation AR-pathway inhibitor (if agent is not listed, must be discussed and approved with CCTG prior to registration). Consult substudies for additional criteria
* Prior cytotoxic therapy: Patients may have received cytotoxic therapy in the castrate sensitive setting as well as up to 1 regimen of cytotoxic therapy in the CRPC setting
* Patients must have an adequate washout prior to enrollment as follows:
* Longest of one of the following:

  * Standard cycle length of standard therapies;
  * Two weeks;
  * The longer of 30 days or 5 half-lives for investigational agents;
* Patients must have discontinued anti-androgens for at least 4 weeks prior to substudy entry/enrollment (at least 6 weeks for bicalutamide).
* LHRH agonist therapy must continue unless surgically castrated. Note: after discussion, CCTG selected patients may be screened prior to adequate washout.
* Patient must have progressed (biochemically or radiologically, as defined in 4.1.4) during or after their last systemic therapy
* Patients must be accessible for treatment and follow up. Patients registered enrolled on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial.
* Investigators must assure themselves the patients enrolled on this trial will be available for complete documentation of the treatment, adverse events, response assessment and follow-up.
* Patients must agree to return to their primary care facility for any adverse events, which may occur through the course of the trial.
* In accordance with CCTG policy, protocol treatment is to begin within 2 working days of patient enrollment.
* Men of childbearing potential must have agreed to use a highly effective contraceptive method during study drug treatment for 6 months after stopping treatment and should not father a child or donate sperm during this period.
* In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation, or vasectomy / vasectomized partner. However, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he is responsible for beginning contraceptive measures.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer, or other solid tumours curatively treated with no evidence of disease for ≥ 2 years.
* Patients with central nervous system (CNS) involvement unless at least 4 weeks from prior therapy completion (including radiation and/or surgery) AND clinically stable and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases. Patients with epilepsy not due to CNS metastases are eligible as long as no contraindication or concern with drug interactions.
* Patients with serious illnesses or medical conditions which could cause unacceptable safety risks or would not permit the patient to be managed according to the protocol. This includes but is not limited to:

  * active infection requiring systemic therapy;
  * active or known human immunodeficiency virus (HIV) with detectable viral load;
  * uncontrolled or recent clinically significant cardiac disease, including:

    * angina pectoris, symptomatic pericarditis, coronary artery bypass grafting, coronary angioplasty, or stenting, or myocardial infarction in the previous 12 months;
    * history of documented congestive heart failure (New York Heart Association functional classification III-IV) or cardiomyopathy;
    * history of any cardiac arrhythmias, e.g. ventricular, supraventricular, nodal arrhythmias, or conduction abnormality in the previous 12 months;
    * patients with uncontrolled hypertension.
  * Patients with significant liver diseases including viral/other hepatitis, current alcohol abuse or cirrhosis.
* Patients who are unable to swallow oral medication and/or have impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g. Crohn's disease, ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, active bowel inflammation (e.g. diverticulitis) or small bowel resection), unless agreed with CCTG (exceptions may be given if parenteral substudy is available/appropriate.
* Patients who require continued or concurrent treatment with:

  * Systemic corticosteroids at a dose equivalent to prednisone > 10 mg daily. Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed.
  * Bisphosphonates / denosumab for reasons other than hypercalcemia, osteoporosis or prevention of skeletal-related events.
  * Other anti-cancer or investigational agents (except LHRH)
* History of hypersensitivity to any of the study drugs or any excipient.
* Patients with a history of non-compliance to medical regimens.
* Patients who have received growth factors within 28 days prior to initiation of dosing of study drug or who are likely to require treatment with growth factors throughout the duration of the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 200 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate defined as proportion of patients who had PSA decline ≥ 50%, complete or partial objective response, or Stable disease for ≥ 12 weeks. | 2 years

SECONDARY OUTCOMES:
Measure effect of each study drug on PSA decline | 2 years
Measure objective response as determined by RECIST 1.1 criteria | 2 years
Number and severity of adverse events | 2 years
Measure effect of each study drug on time to PSA progression | 2 years
To summarize progression-free survival | 2 years
To summarize overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kolinsky, Study Chair — Cross Cancer Institute, Edmonton, AB Canada; Som Mukherjee, Study Chair — Juravinski Cancer Centre at Hamilton Health Sciences Centre, ON Canada; Michael Ong, Study Chair — Ottawa Hospital Research Institute, Ottawa, ON Canada; Kim Chi, Study Chair — BCCA - Vancouver Cancer Centre; Aaron Hansen, Study Chair — University Health Network, Toronto, ON, Canada; Sebastien Hotte, Study Chair — Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, ON Canada; Zineb Hamilou, Study Chair — CHUM-Centre Hospitalier de l'Universite de Montreal
Locations (11):
- Canada (11):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maia MC, Salgia M, Pal SK. Harnessing cell-free DNA: plasma circulating tumour DNA for liquid biopsy in genitourinary cancers. Nat Rev Urol. 2020 May;17(5):271-291. doi: 10.1038/s41585-020-0297-9. Epub 2020 Mar 17. PMID 32203306